CLINICAL TRIAL: NCT04923893
Title: A Phase 3 Randomized Study Comparing Bortezomib, Lenalidomide and Dexamethasone (VRd) Followed by Ciltacabtagene Autoleucel, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against BCMA Versus Bortezomib, Lenalidomide, and Dexamethasone (VRd) Followed by Lenalidomide and Dexamethasone (Rd) Therapy in Participants With Newly Diagnosed Multiple Myeloma for Whom Hematopoietic Stem Cell Transplant is Not Planned as Initial Therapy
Brief Title: A Study of Bortezomib, Lenalidomide and Dexamethasone (VRd) Followed by Cilta-cel, a CAR-T Therapy Directed Against BCMA Versus VRd Followed by Lenalidomide and Dexamethasone (Rd) Therapy in Participants With Newly Diagnosed Multiple Myeloma for Whom ASCT is Not Planned as Initial Therapy
Acronym: CARTITUDE-5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109015; 68284528MMY3004 (Other: Janssen Research & Development, LLC); 2021-001242-35 (EudraCT Number); 2023-505850-16-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05346835 (Available)
Record Dates: First submitted 2021-06-10; First posted 2021-06-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed Multiple Myeloma; Cellular Therapy; CAR-T Therapy; BCMA CAR-T
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Lenalidomide; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: VRd+Rd (Standard Therapy) (Experimental): Participants will receive bortezomib, lenalidomide, and dexamethasone (VRd) regimen for 6 cycles before randomization. Following randomization, participants in Arm A will receive 2 more cycles of VRd. In VRd treatment, participants will receive bortezomib 1.3 milligram per meter square (mg/m^2) subcutaneously (SC) on Days 1, 4, 8 and 11 of each cycle (Cycles 1 to 8), oral lenalidomide 25 mg on Days 1 to 14 of each cycle (Cycles 1 to 8) and oral dexamethasone 20 mg on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each cycle (Cycles 1 to 8). Each cycle will consist of 21 days. After 8 cycles of VRd, treatment will continue with lenalidomide and dexamethasone (Rd) maintenance therapy. In Rd treatment, participants will receive oral lenalidomide 25 mg on Days 1 to 21 of each cycle and oral dexamethasone 40 mg on Days 1, 8, 15, and 22 of each cycle. Each cycle will consist of 28 days. Participants will continue to receive Rd until confirmed progressive disease or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Lenalidomide
- Arm B: VRd+Ciltacabtagene Autoleucel (Cilta-cel) (Experimental): Participants will receive VRd regimen for 6 cycles before randomization. Following randomization, participants in Arm B will undergo apheresis and receive two more cycles of VRd as bridging therapy. In VRd treatment, participants will receive bortezomib 1.3 mg/m^2 SC on Days 1, 4, 8 and 11 of each cycle for Cycles 1 to 8; oral lenalidomide 25 mg on days 1 to 14 of each cycle for Cycles 1 to 8 and oral dexamethasone 20 mg on days 1, 2, 4, 5, 8, 9, 11 and 12 of each cycle for Cycles 1 to 8. Each cycle will consist of 21 days. After 8 cycles of VRd, participants will receive a conditioning regimen (cyclophosphamide 300 mg/m^2 intravenous [IV] and fludarabine 30 mg/m^2 IV daily for 3 days) and Cilta-cel infusion 0.75*10^6 chimeric antigen receptor (CAR)-positive viable T cells/kilogram (kg).
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Cilta-cel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be administered SC.
Drug: Dexamethasone — Dexamethasone will be administered orally.
Drug: Lenalidomide — Lenalidomide will be administered orally.
Drug: Cilta-cel — Cilta-cel infusion will be administered.
  Other Names: JNJ-68284528
  Arms: Arm B: VRd+Ciltacabtagene Autoleucel (Cilta-cel)
Drug: Cyclophosphamide — Cyclophosphamide will be administered intravenously.
  Arms: Arm B: VRd+Ciltacabtagene Autoleucel (Cilta-cel)
Drug: Fludarabine — Fludarabine will be administered intravenously.
  Arms: Arm B: VRd+Ciltacabtagene Autoleucel (Cilta-cel)

SUMMARY:
The purpose of this study is to compare the efficacy of Bortezomib, Lenalidomide and Dexamethasone (VRd) induction followed by a single administration of ciltacabtagene autoleucel (cilta-cel) versus VRd induction followed by Lenalidomide and Dexamethasone (Rd) maintenance in newly diagnosed multiple myeloma participants for whom ASCT is not planned as initial therapy in terms of Progression Free Survival (PFS).

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant plasma cell disorder characterized by the production of monoclonal immunoglobulin (Ig) proteins or protein fragments (M proteins) that have lost their function. JNJ-68284528 (ciltacabtagene autoleucel [cilta-cel]) is an autologous chimeric antigen receptor T cell (CAR-T) therapy that targets B-cell maturation antigen (BCMA), a molecule expressed on the surface of mature B lymphocytes and malignant plasma cells. The primary hypothesis of this study is that in participants with newly diagnosed MM, treatment with VRd induction followed by a single administration of cilta-cel will significantly improve progression free survival compared to Bortezomib, Lenalidomide and Dexamethasone (VRd) induction followed by Rd maintenance. The study will screen participants with newly diagnosed MM who are not planned to receive autologous stem cell transplant (ASCT) as initial therapy. This study will be conducted in 4 phases: Screening (up to 28 days), Pre-randomization Treatment, Treatment, and Follow-up. Assessments like patient-reported outcome(s) (PROs), electrocardiogram (ECG), vital signs and pharmacokinetics will be performed during the study. Safety evaluations will include review of adverse events, laboratory test results, vital sign measurements, physical examination findings, assessment of cardiac function, Immune-Effector Cell-Associated Encephalopathy (ICE) and handwriting assessments (only for Arm B) and Eastern Cooperative Oncology Group (ECOG) performance status. Safety data will be periodically reviewed by an Independent Data Monitoring Committee (IDMC). The duration of the study is approximately 12 years 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma (MM) according to International Myeloma Working Group (IMWG) diagnostic criteria
* Measurable disease at screening as defined by any of the following: Serum monoclonal paraprotein (M-protein) level greater than or equal to (>=)1.0 gram per deciliter (g/dL) or urine M-protein level >=200 milligram (mg)/24 hours; or Light chain MM in whom only measurable disease is by serum free light chain (FLC) levels: Serum immunoglobin (Ig) free light chain >=10 milligrams per deciliter (mg/dL) and abnormal serum Ig kappa/lambda FLC ratio
* Eastern Cooperative Oncology Group Performance Status grade of 0 or 1
* Not considered for high-dose chemotherapy with Autologous Stem Cell Transplant (ASCT) due to: Ineligible due to advanced age; or Ineligible due to presence of comorbid condition(s) likely to have a negative impact on tolerability of high-dose chemotherapy with ASCT; or Deferral of high-dose chemotherapy with ASCT as initial treatment
* A woman of childbearing potential (WOCBP) must have 2 negative highly sensitive serum or urine pregnancy tests (beta-human chorionic gonadotropin) prior to starting Bortezomib, Lenalidomide and Dexamethasone (VRd) and must agree to further testing during the study.
* Clinical laboratory values meeting the following criteria during the screening phase: hemoglobin greater than or equal to (>=) 8.0 g/dL (>=5 millimoles per liter [mmol/L]), recombinant human erythropoietin use is permitted; platelets >=75 *10^9/L; absolute lymphocyte count >=0.3 *10^9/L; absolute neutrophil count (ANC) >=1.0 ×10^9/L (prior growth factor support is permitted but must be without support in the 7 days prior to the laboratory test); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to (<=) 3.0 * upper limit of normal (ULN); estimated glomerular filtration rate >=40 milliliter per minute/1.73 meter square (mL/min/1.73 m^2) based upon modified diet in renal disease formula (MDRD-4) calculation or a 24-hour urine collection; total bilirubin <=2.0 * ULN; except in participants with congenital hyperbilirubinemia, such as Gilbert syndrome (in which case direct bilirubin <=2.0 * ULN is required)

Exclusion Criteria:

* Frailty index of >=2 according to Myeloma Geriatric Assessment score
* Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5
* Known active, or prior history of central nervous system (CNS) involvement or clinical signs of meningeal involvement of MM
* Stroke or seizure within 6 months of signing Informed Consent Form (ICF)
* Seropositive for human immunodeficiency virus (HIV)
* Vaccinated with live, attenuated vaccine within 4 weeks prior to first dose of VRd
* Participant must not require continuous supplemental oxygen
* Hepatitis B infection
* Hepatitis C infection
* Prior treatment with chimeric antigen receptor T (CAR-T) therapy directed at any target
* Any therapy that is targeted to B-cell maturation antigen (BCMA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2029-02-14 (Estimated); Study Completion 2036-09-22 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 4 years and 5 months
  Progression-free survival is defined as the time from the date of randomization to the date of first documented Progressive Disease (PD), as defined in the International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Sustained Minimal Residual Disease (MRD) Negative CR | Up to 12 years and 5 months
  Sustained MRD negative complete response (CR) as determined by next generation sequencing (NGS) with sensitivity of 10^-5, and defined by MRD negative CR plus at least 12 months durability of the MRD negative CR status.
MRD Negative CR at 9 Months | 9 months
  MRD negative CR rate at 9 months is defined as the percentage of participants who achieve MRD negative CR status at 9±3 months after the randomization date.
Overall MRD Negative CR | Up to 12 years and 5 months
  Overall MRD negative is defined as the percentage of participants who achieve MRD negativity at any time after the date of randomization before initiation of subsequent therapy.
Overall Survival (OS) | Up to 12 years and 5 months
  Overall survival is measured from the date of randomization to the date of the participant's death.
Complete Response or Better | Up to 12 years and 5 months
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response according to the IMWG criteria.
Time to Subsequent Anti-myeloma Therapy | Up to 12 years and 5 months
  Time to subsequent anti-myeloma therapy is defined as the time from randomization to the start of subsequent anti-myeloma therapy.
Progression Free Survival on Next-line Therapy (PFS2) | Up to 12 years and 5 months
  PFS2 is defined as the time interval between the date of randomization and date of event, which is defined as PD as assessed by investigator that starts after the next line of subsequent therapy, or death from any cause, whichever occurs first.
Number of Participants with Adverse Events (AEs), Abnormalities in Laboratory Parameters, 12-Lead Electrocardiogram (ECG), Physical Examination, and Vital Signs | Up to 12 years and 5 months
  Number of participants with AEs, abnormalities in laboratory parameters (complete blood count [CBC] with differential, coagulation, chimeric antigen receptor T cell [CAR-T] chemistry, full metabolic panel etc.), 12-lead ECG, physical examination, and vital signs will be reported.
Arm B: Systemic Cytokine Concentrations | Up to Day 112
  Serum or plasma proteomic profiling of cytokines (such as interleukin [IL] 6, IL-15, and IL 10) concentrations will be measured for biomarker assessment.
Arm B: Levels of Chimeric Antigen Receptor T cell (CAR-T) Cell Activation Markers | Up to 12 years and 5 months
  CAR-T cell activation markers including, but not limited to, CD4+, CD8+, CD25+, central memory, effector memory cells will be reported. An evaluation of cell populations may be performed by flow cytometry, cytometry by time of flight (CyTOF), single cell RNA sequencing (scRNAseq) or similar technologies and be correlated with response.
Arm B: Levels of Soluble B-cell Maturation Antigen (BCMA) | Up to 1 year
  Levels of soluble BCMA will be reported.
Arm B: Levels of Cilta-cel Expansion (proliferation), and Persistence | Up to 12 years and 5 months
  Levels of cilta-cel expansion (proliferation), and persistence via monitoring CAR-T positive cell counts and CAR transgene level will be reported.
Arm B: Number of Participants with Anti-cilta-cel Antibodies | Up to 12 years and 5 months
  Number of participants with anti-cilta-cel antibodies will be reported.
Arm B: Number of Participants with Presence of Replication Competent Lentivirus | Up to 12 years and 5 months
  Number of participants with presence of replication competent lentivirus will be reported.
Change from Baseline in Health-Related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) Scale Score | Baseline up to 12 years and 5 months
  The EORTC QLQ-C30 includes 30 items in 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The responses are reported using a verbal rating scale. The item and scale scores are transformed to a 0 to 100 scale. A higher score represents greater HRQoL, better functioning, and more (worse) symptoms.
Change from Baseline in Health-Related Quality of Life as Assessed by MySIm-Q Scale Score | Baseline up to 12 years and 5 months
  The MySIm-Q is a disease-specific PRO assessment complementary to the EORTC-QLQ-C30. It includes 17 items with recall period of "7 days" and responses are reported on a 5-point verbal rating scale. Item responses are scored from 0 to 4. Higher scores indicate greater severity/impact.
Change from Baseline in Health-Related Quality of Life as Assessed by European Quality of Life - 5 Dimensions-5 Levels (EQ-5D-5L) Scale Score | Baseline up to 12 years and 5 months
  The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems, where Level 1: no problem, Level 2: slight problems, Level 3: moderate problems, Level 4: severe problems and Level 5: extreme problems, plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in Health-Related Quality of Life as Assessed by Patient Global Impression of Symptom Severity (PGIS) Scale Score | Baseline up to 12 years and 5 months
  The PGIS uses 2 items to assess the participant's perception of the severity of their disease symptoms and impact using a 5-point verbal rating scale. Score ranges from 1 (None) to 5 (Very Severe).
Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Items | Up to 161 days
  The National Cancer Institute's PRO-CTCAE is an item library of common adverse events experienced by people with cancer that are appropriate for self-reporting. Each symptom selected for inclusion can be rated by up to 3 attributes characterizing the presence/frequency, severity, and/or interference that ranges from 0 to 4 with higher scores indicating higher frequency or greater severity/impact.
Time to Worsening of Symptoms, Functioning and Overall Well-being | Up to 12 year and 5 months
  Time to worsening is measured as the interval from the date of randomization to the start date of worsening in MySIm-Q symptom, impact, or total scores.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (136):
- United States (19):
  - UCSF, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami Health System, Miami, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - University Of Maryland Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian-Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Aleman, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Privado Universitario De Cordoba, Córdoba
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown
  - St Vincents Hospital Melbourne, Fitzroy
  - Austin Health, Heidelberg
  - Royal Brisbane and Womens Hospital, Herston
  - Alfred Health, Melbourne
  - Peter MacCallum Cancer Centre, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Calvary Mater Newcastle Hospital, Waratah
  - Western Sydney Local Health District, Westmead
- Austria (4):
  - Medizinische Universitat Graz, LKH-Univ.Klinikum Graz, Klinische Abteilung für Hämatologie, Graz
  - Krankenhaus der Elisabethinen Linz, Linz
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medical University of Vienna Universitatsklinik fur Innere Medizin I, Vienna
- Belgium (5):
  - Universitair Ziekenhuis - Antwerpen, Antwerp
  - AZ St.-Jan Brugge-Oostende AV, Bruges
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
- Brazil (3):
  - Hospital Sao Rafael, Salvador
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Canada (5):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (3):
  - Aarhus University Hospital, Aarhus C
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense C
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku
- France (5):
  - Centre Hospitalier Régional Universitaire de Lille, Hôpital Claude Huriez, Lille
  - C.H.U. Hotel Dieu - France, Nantes
  - Hopital Saint Louis, Paris
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - Institut Universitaire du cancer de Toulouse-Oncopole, Toulouse
- Germany (11):
  - Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Klinikum Großhadern der Ludwig-Maximilians-Universität, München
  - Universitaetsklinikum Regensburg, Regensburg
  - Klinikum der Eberhard Karls Universitaet Abt fur innere Med II Haematologie Onkologie Germany, Tübingen
  - Universitatsklinikum Wurzburg, Würzburg
- Greece (3):
  - Alexandra General Hospital of Athens, Athens
  - Attikon University General Hospital of Attica, Athens
  - G.Papanikolaou, Thessaloniki
- Hungary (2):
  - Del Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet Szent Laszlo Telephely, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- St James Hospital, Dublin, Ireland
- Israel (3):
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Sheba Medical Center Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (10):
  - Juntendo University Hospital, Bunkyō City
  - Kyushu University Hospital, Fukuoka
  - Hyogo Medical University Hospital, Hyôgo
  - Kanazawa University Hospital, Kanazawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Nagoya City University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Japanese Red Cross Medical Center, Shibuya City
- Netherlands (4):
  - VU Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - UMC Radboud, Nijmegen
  - Erasmus MC, Rotterdam
- Oslo universitetssykehus HF, Rikshospitalet, Oslo, Norway
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut BadawczyOddz w Gliwicach, Gliwice
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Portugal (2):
  - Instituto Portugues de Oncologia, Lisbon
  - Instituto Portugues de Oncologia, Porto
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (11):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Instituto Catalan Deoncologia Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Virgen de La Arrixaca, Murcia
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Universitetssjukhuset, Linköping
  - Skane University Hospital, Lund
- Switzerland (3):
  - Universitatsspital Basel, Basel
  - Inselspital Universitatsspital Bern, Bern
  - Kantonsspital St Gallen, Sankt Gallen
- United Kingdom (7):
  - University Hospitals Birmingham NHS Trust,, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University College Hospital, London
  - Kings College Hospital, London
  - Manchester Royal Infirmary, Manchester
  - The Royal Marsden NHS Trust Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- See also: Click here to learn more about the 68284528MMY3004 (CARTITUDE-5) trial (US only) — https://sparkcures.com/trial/1182/nct04923893?utm_source=ctgov&utm_medium=organic&utm_campaign=cartitude5